CLINICAL TRIAL: NCT02152969
Title: An Open-label, Multiple-dose, Two-arm Clinical Study to Evaluate the Drug-drug Interaction and Safety of Telmisartan, Amlodipine and/or Chlorthalidone in Healthy Adult Volunteers
Brief Title: Drug-drug Interaction Study (Telmisartan, Amlodipine, Chlorthalidone)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: YH22162-101
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Amlodipine; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part B (Other): Arm to evaluate influence of Chlorthalidone on pharmacokinetics of amlodipine and telmisartan.
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Chlorthalidone
- Part A (Other): Arm to evaluate influence of amlodipine and telmisartan on pharmacokinetics of Chlorthalidone.
  Interventions: Drug: Telmisartan; Drug: Amlodipine; Drug: Chlorthalidone

INTERVENTIONS:
Drug: Telmisartan
Drug: Amlodipine
Drug: Chlorthalidone

SUMMARY:
To evaluate Drug-drug interaction

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Drug-Drug(telmisartan, amlodipine and/ or chlorthalidone) interaction and safety in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Participant who has a body weight that is ≥55kg(male) or ≥50kg(female) with ideal body weight of 80-120% (ideal body weight)
2. Who has not suffered from clinically significant disease
3. Provision of signed written informed consent

Exclusion Criteria:

1. History of and clinically significant disease psychiatric, or malignancy.
2. A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs.
3. Administration of other investigational products within 3 months prior to the first dosing.
4. Administration of herbal medicine within 2 weeks or administration of ethical drugs within 2 weeks or administration of over-the-counter (OTC) drugs within 1 week prior to the first dosing of the investigational product (if the investigator (study doctor) determines that the person meets other criteria appropriately, the relevant person may participate in the study).
5. Volunteers considered not eligible for the clinical trial by the investigator (study doctor) due to reasons including laboratory test results, ECGs, or vital signs.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
AUCt ss, Cmax ss of telmisartan/amlodipine/chlorthalidone | Totally 28points for 24 hours

SECONDARY OUTCOMES:
Cmin ss, tmax ss, t1/2 of telmisartan/amlodipine/chlorthalidone | Totally 28points for 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dong Seok Yim, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea Seoul St.Mary's Hospital, Seoul, South Korea